CLINICAL TRIAL: NCT02015819
Title: A Phase I Study of Cytosine Deaminase-Expressing Neural Stem Cells in Combination With Oral 5-Fluorocytosine and Leucovorin for the Treatment of Recurrent High-Grade Gliomas
Brief Title: Genetically Modified Neural Stem Cells, Flucytosine, and Leucovorin for Treating Patients With Recurrent High-Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13401; NCI-2013-02346 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13401 (Other: City of Hope Medical Center); FD-R-004816 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor; Anaplastic Oligoastrocytoma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Flucytosine; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (neural stem cells, flucytosine, leucovorin) (Experimental): Patients receive CD-expressing neural stem cells intracranially on days 1 and 15. Flucytosine is taken orally every 6 hours on days 4-10 and 18-24. Depending on when a subject enters the study, they may also be given leucovorin orally every 6 hours on days 4-10 and 18-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Dose escalation used the following dose levels:
  Dose Level 1 (NSC 5x10^7 and 5-FC 37.5 mg/kg)
  Dose Level 2 (NSC 1x10^8 and 5-FC 37.5 mg/kg)
  Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg)
  Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis
  Interventions: Biological: E. coli CD-expressing genetically modified neural stem cells; Drug: flucytosine; Drug: leucovorin calcium; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: E. coli CD-expressing genetically modified neural stem cells — Given intracranially
  Other Names: HB1.F3.CD neural stem cells
Drug: flucytosine — Given orally
  Other Names: 5-FC; 5-fluorocytosine; Ro 2-9915
Drug: leucovorin calcium — Given orally
  Other Names: CF; CFR; LV
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and determines the best dose of genetically modified neural stem cells and flucytosine when given together with leucovorin for treating patients with recurrent high-grade gliomas. Neural stem cells can travel to sites of tumor in the brain. The neural stem cells that are being used in this study were genetically modified express the enzyme cytosine deaminase (CD), which converts the prodrug flucytosine (5-FC) into the chemotherapy agent 5-fluorouracil (5-FU). Leucovorin may help 5-FU kill more tumor cells. The CD-expressing neural stem cells are administered directly into the brain. After giving the neural stem cells a few days to spread out and migrate to tumor cells, research participants take a 7 day course of oral 5-FC. (Depending on when a research participant enters the study, they may also be given leucovorin to take with the 5-FC.) When the 5-FC crosses into brain, the neural stem cells convert it into 5-FU, which diffuses out of the neural stem cells to preferentially kill rapidly dividing tumor cells while minimizing toxicity to healthy tissues. A Rickham catheter, placed at the time of surgery, will be used to administer additional doses of NSCs every two weeks, followed each time by a 7 day course of oral 5-FC (and possibly leucovorin). This neural stem cell-based anti-cancer strategy may be an effective treatment for high-grade gliomas.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the phase II recommended dose of intracerebrally administered cytosine deaminase (CD)-expressing neural stem cells (NSCs) in combination with oral 5-fluorocytosine (FC) (flucytosine) and leucovorin.

II. To determine the feasibility of treating study patients with more than 1 dose of NSCs followed by 7-day courses of 5-FC and leucovorin.

SECONDARY OBJECTIVES:

I. To assess for possible development of NSC immunogenicity (anti-NSC T cell and/or antibody response) with repeat doses of NSCs.

II. To characterize the relationship between intracerebral and systemic concentrations of 5-FC and 5-FU at the maximum tolerated dose/maximum feasible dose level.

III. To describe the clinical benefit (defined as stable disease, partial response, or complete response) of this treatment regimen.

IV. To determine, at time of autopsy, the fate of the NSCs.

OUTLINE: This is dose-escalation study of CD-expressing genetically modified neural stem cells and flucytosine.

Patients receive CD-expressing neural stem cells intracranially (IC) on days 1 and 15 and flucytosine orally (PO) every 6 hours on days 4-10 and 18-24. Depending on when a subject enters the study, they may also be given leucovorin orally every 6 hours on days 4-10 and 18-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 30 days, 3 months, 6 months, 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient has had a prior, histologically-confirmed, diagnosis of a grade III or IV glioma (including glioblastoma, anaplastic oligodendroglioma, or anaplastic astrocytoma, gliosarcoma, anaplastic oligodendroglioma, or anaplastic oligoastrocytoma), or has a prior, histologically-confirmed, diagnosis of a grade II glioma and now has radiographic findings consistent with a high-grade glioma (grade III or IV)
* Imaging studies show evidence of recurrent, supratentorial tumor(s). The presence of infratentorial tumor is allowed as long as the patient also has supratentorial disease that is amenable to resection or biopsy.
* Patient's high-grade glioma has recurred or progressed after prior treatment with brain radiation and temozolomide
* Patient has a Karnofsky performance status of >= 70%
* Patient has a life expectancy of >= 3 months
* Female patients of childbearing potential and sexually-active male patients must agree to use an effective method of contraception while participating in this study; women of childbearing potential must have a negative pregnancy test =< 2 weeks prior to registration
* The patient must be in need of a craniotomy for tumor resection or a stereotactic brain biopsy for the purpose of diagnosis or differentiating between tumor progression versus treatment-induced effects following radiation therapy +/- chemotherapy
* Based on the neurosurgeon's judgement, there is no anticipated physical connection between the post-resection tumor cavity and the cerebral ventricles
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3
* Platelet count >= 100,000 cells/mm^3
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 4 times the institutional upper limit of normal
* Serum creatinine =< the institutional upper limit of normal
* There is no limit to the number of prior therapies
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patient has anti-human leukocyte antigen (HLA) antibodies specific for HLA antigens expressed by the NSCs
* Patient has not recovered from any toxicity of prior therapies; an interval of

  * At least 6 weeks must have elapsed since taking a nitrosourea-containing chemotherapy regimen
  * At least 4 weeks since completing a non-nitrosourea-containing cytotoxic chemotherapy regimen (except temozolomide: only an interval of 23 days is required from the last dose administered when patient has been recently treated with the standard temozolomide regimen of daily for 5 days, repeated every 28 days)
  * At least 2 weeks from taking the last dose of targeted agent
  * At least 4 weeks from the last dose of bevacizumab
* Patient is unable to undergo a magnetic resonance imaging (MRI)
* Patient is allergic to 5-FC, leucovorin, or 5-FU
* Patient has chronic or active viral infections of the central nervous system (CNS)
* Patient has a coagulopathy or bleeding disorder
* Patient has an uncontrolled illness including ongoing or active infection
* Patient is receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* Patient has had prior therapy with neural stem cells
* Patient is pregnant or breast feeding; pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is participating in this study
* Patient has another active malignancy
* Non-compliance; a patient has a serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the safety monitoring requirements and completion of treatment according to this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2017-10-07 (Actual); Study Completion 2017-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jana Portnow, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 (NSC 5x10^7 and 5-FC 37.5 mg/kg); Dose Level 2 (NSC 1x10^8 and 5-FC 37.5 mg/kg); Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg): Patients receive CD-expressing neural stem cells intracranially on days 1 and 15. Flucytosine is taken orally every 6 hours on days 4-10 and 18-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis: Patients receive CD-expressing neural stem cells intracranially on days 1 and 15. Flucytosine is taken orally every 6 hours on days 4-10 and 18-24. They will also be given leucovorin orally every 6 hours on days 4-10 and 18-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level 1 (NSC 5x10^7 and 5-FC 37.5 mg/kg) | Dose Level 2 (NSC 1x10^8 and 5-FC 37.5 mg/kg) | Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis
Started | 3 | 3 | 3 | 7
Completed | 3 | 3 | 3 | 6
Not Completed | 0 | 0 | 0 | 1
Not completed — Rickham catheter was misaligned | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis: Patients receive CD-expressing neural stem cells intracranially on days 1 and 15. Flucytosine is taken orally every 6 hours on days 4-10 and 18-24. Leucovorin orally every 6 hours on days 4-10 and 18-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 (NSC 5x10^7 and 5-FC 37.5 mg/kg) | Dose Level 2 (NSC 1x10^8 and 5-FC 37.5 mg/kg) | Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis | Total
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 16
Age, Continuous [Median (Full Range); unit: years] | 59 [48 to 59] | 40 [26 to 64] | 57 [54 to 65] | 58 [45 to 71] | 57 [26 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 3
  Male | 1 | 3 | 2 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 3 | 3 | 1 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 2 | 2 | 3 | 7 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) and Maximum Tolerated Dose (MTD)
Description: Number of DLTs per dose level and the MTD/MFD.
Time Frame: Day 28 of course 1
Population: 1 participant in dose level 4 was unevaluable and had to be replaced after receiving the first dose of CD-NSCs due to the tip of the Rickham catheter migrating into the lateral ventricle.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: (NSC 5x10^7 and 5-FC 37.5 mg/kg); Dose Level 2: (NSC 1x10^8 and 5-FC 37.5 mg/kg); Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg); Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg + Leucovorin + Microdialysis: Patients receive CD-expressing neural stem cells intracranially on days 1 and 15. Flucytosine is taken orally every 6 hours on days 4-10 and 18-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level 1: (NSC 5x10^7 and 5-FC 37.5 mg/kg) | Dose Level 2: (NSC 1x10^8 and 5-FC 37.5 mg/kg) | Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg + Leucovorin + Microdialysis
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Dose Level 1: (NSC 5x10^7 and 5-FC 37.5 mg/kg) vs Dose Level 2: (NSC 1x10^8 and 5-FC 37.5 mg/kg) vs Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) vs Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg + Leucovorin + Microdialysis; Test type: Other; MFD was determined to be 1.5x10^8 in combination with oral 5-FC 37.5 mg/kg and leucovorin 25 mg every 6 hours for 7 days

2. Primary Outcome: Number of Participants With Mechanical Issues With Repeat Administrations of NSCs Via Rickham
Description: Number of participants with mechanical issues with repeat administrations of NSCs via Rickham.
Time Frame: 28 days after last infusion of NSCs, up to 6 months total
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (NSC 5x10^7 and 5-FC 37.5 mg/kg) | Dose Level 2 (NSC 1x10^8 and 5-FC 37.5 mg/kg) | Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis
Number analyzed (Participants) | 3 | 3 | 3 | 7
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Developing Antibodies Against NSCs
Description: Development of a antibody response to the NSCs will be evaluated by flow cytometry. Data from assessing for possible development of NSC immunogenicity with repeat exposure will be presented in an exploratory fashion using descriptive statistics.
Time Frame: While receiving treatment, up to 6 months.
Population: 2 participants in dose level 4 were not assessed in this analysis because one participant only received one dose of CD-NSCs and the other we were unable to obtain post second CD-NSC dose serum sample to analyze.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (NSC 5x10^7 and 5-FC 37.5 mg/kg) | Dose Level 2 (NSC 1x10^8 and 5-FC 37.5 mg/kg) | Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis
Number analyzed (Participants) | 3 | 3 | 3 | 5
Participants | 0 | 2 | 0 | 1

4. Secondary Outcome: Average Steady State Levels of 5-FC and 5-FU in the Brain
Description: Pharmacokinetic (PK) data from the patients who undergo intracerebral microdialysis (dose level 4) will be summarized using descriptive statistics. All summaries will be exploratory in spirit.
Time Frame: Following the first dose of 5-FC, samples were collected every hour for 24 hours and then every 3 hours thereafter until the end of the 7-day course of 5-FC or until the microdialysis catheter stopped functioning.
Population: Only participants in dose level 4 received intracerebral microdialysis and are included in this analysis
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis
Number analyzed (Participants) | 7
µmol/L
  average steady state levels of 5-FC in the brain | 213 (58)
  average steady state levels of 5-FU in the brain | 0.03 (0.01)

5. Secondary Outcome: Average Steady State Levels of 5-FC Concentrations in Plasma
Description: PK data from the patients who undergo intracerebral microdialysis (dose level 4) will be summarized using descriptive statistics.
Time Frame: Samples were obtained prior to the first dose of 5-FC then every 30 minutes for 3 hours, additional samples at 4 and 6 hours after the morning doses on days 4, 5. On days 6, 7, 8 blood samples were collected just before morning dose and 90 minutes later
Population: Only participants in dose level 4 received intracerebral microdialysis and are included in this analysis
Measure: Mean (Standard Error); unit: µmol/L
Arm/Group | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis
Number analyzed (Participants) | 7
µmol/L | 748 (218)

6. Secondary Outcome: Comparison of 5-FC in the Brain to 5-FC in the Plasma
Description: PK data from the patients who undergo intracerebral microdialysis (dose level 4) will be summarized using the mean ratio of average brain interstitial 5-FC concentrations to the average steady-state plasma levels.
Time Frame: The ratio of average brain interstitial 5-FC and 5-FU concentrations to average plasma steady-state levels was calculated using all measured data.
Population: Only participants in dose level 4 received intracerebral microdialysis and are included in this analysis
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis
Number analyzed (Participants) | 7
ratio | 29 (21)

7. Secondary Outcome: Summary of Tumor Response Using the Response Assessment in Neuro-Oncology (RANO) Criteria
Description: Per RANO criteria:
  Complete Response (CR): Complete disappearance of all enhancing disease that is sustained for at least 4 weeks, stable or improved non-enhancing FLAIR/T2 lesions, no new lesions, off corticosteroids, and neurologically stable or improved.
  Partial Response (PR): >= 50% decrease of all measurable enhancing lesions, sustained or at least 4 weeks, no progression of non-measurable disease, stable or improved non-enhancing FLAIR/T2 lesions, non new lesions, corticosteroid dose stable or reduced, and neurologically stable or improved.
  Stable Disease (SD): Dose not qualify for CR, PR, or PD, stable non-enhancing FLAIR/T2 lesions, stable or reduced corticosteroids, clinically stable.
  Progressive Disease (PD): >=25% increase in enhancing lesion despite stable or increasing steroid dose, increase (significant) in non-enhancing T2/FLAIR lesions that is not attributable to other non-tumor causes, any new lesions, clinical deterioration
Time Frame: Up to 3 years post NSC infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (NSC 5x10^7 and 5-FC 37.5 mg/kg) | Dose Level 2 (NSC 1x10^8 and 5-FC 37.5 mg/kg) | Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis
Number analyzed (Participants) | 3 | 3 | 3 | 7
Participants
  Stable Disease | 2 | 0 | 0 | 1
  Progressive Disease | 1 | 3 | 3 | 4
  Ineligible for Disease Response | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: During and after treatment, up to 20 months
Arm/Group | Dose Level 1 (NSC 5x10^7 and 5-FC 37.5 mg/kg) | Dose Level 2 (NSC 1x10^8 and 5-FC 37.5 mg/kg) | Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 7/7
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/3 | 4/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (NSC 5x10^7 and 5-FC 37.5 mg/kg) (N=3) | Dose Level 2 (NSC 1x10^8 and 5-FC 37.5 mg/kg) (N=3) | Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) (N=3) | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis (N=7)
Seizure (Nervous system disorders) | 1 | 0 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 1 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (NSC 5x10^7 and 5-FC 37.5 mg/kg) (N=3) | Dose Level 2 (NSC 1x10^8 and 5-FC 37.5 mg/kg) (N=3) | Dose Level 3 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) (N=3) | Dose Level 4 (NSC 1.5x10^8 and 5-FC 37.5 mg/kg) + Leucovorin + Microdialysis (N=7)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 6
Sinus bradycardia (Cardiac disorders) | 2 | 1 | 0 | 4
Sinus tachycardia (Cardiac disorders) | 2 | 2 | 1 | 4
Premature ventricular contractions (Cardiac disorders) | 1 | 0 | 0 | 0
tachypnea (Cardiac disorders) | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 2 | 0 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 1 | 0 | 0
Floaters (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 5
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 1
Ulceration on Tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0
mouth sores (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 1 | 0
Edema face (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 1 | 4
Fever (General disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 2 | 1 | 2 | 5
Pain (General disorders) | 1 | 2 | 1 | 6
Edema limbs (General disorders) | 2 | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 1 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 3
numbness at surgical site (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
swelling, right side of forehead (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0
Cholesterol high (Investigations) | 1 | 0 | 0 | 0
INR increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 1 | 2 | 6
Platelet count decreased (Investigations) | 2 | 1 | 2 | 7
Weight gain (Investigations) | 2 | 1 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 2
White blood cell decreased (Investigations) | 1 | 0 | 0 | 2
Hemoglobin increased (Investigations) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 6
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 3
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 1
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 1 | 3
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 3 | 5
Concentration impairment (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 2 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 2 | 3
Headache (Nervous system disorders) | 3 | 3 | 3 | 7
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 2
Lethargy (Nervous system disorders) | 0 | 1 | 1 | 3
Memory impairment (Nervous system disorders) | 1 | 2 | 2 | 4
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0 | 1 | 2
Seizure (Nervous system disorders) | 2 | 2 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 3
Spasticity (Nervous system disorders) | 1 | 1 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 1 | 2
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 2
Left-sided balance/coordination problems (Nervous system disorders) | 1 | 0 | 0 | 0
aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
hygroma (Nervous system disorders) | 0 | 0 | 0 | 1
tightness/swelling at right side of brain (Nervous system disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 3 | 3
Confusion (Psychiatric disorders) | 2 | 1 | 2 | 4
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 2
Emotional lability (Psychiatric disorders) | 0 | 0 | 1 | 0
MOOD CHANGES (Psychiatric disorders) | 0 | 1 | 0 | 0
frustration (Psychiatric disorders) | 1 | 0 | 0 | 0
impulsive (Psychiatric disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 3
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
Lung congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin sore (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
blisters (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
excoriation / rash at coccyx (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 3 | 2 | 6
Hypotension (Vascular disorders) | 3 | 0 | 2 | 2
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT02015819/Prot_SAP_000.pdf